CLINICAL TRIAL: NCT01937208
Title: A Prospective, Randomised Phase 3 Study of High-dose Versus Standard-dose Radiation of Inoperable Esophageal Carcinoma Treated With Concurrent Chemoradiation
Brief Title: Comparable Study of Different Radiation Dose in Esophageal Carcinoma
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ESC-130825
Record Dates: First submitted 2013-08-25; First posted 2013-09-09 (Estimated); Last update posted 2013-09-09 (Estimated); Status verified 2013-09

CONDITIONS: Esophageal Carcinoma
Keywords: Esophageal Carcinoma; chemoradiation; radiation dose
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Radiotherapy, Intensity-Modulated; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- high-dose (Experimental): concurrent chemoradiation:CT:DDP 25mg/m2 D1+docetaxel 25mg/m2 D1,Weekly for 5 wks;RT：60Gy/30F/6W(3D-CRT or IMRT).Then,2 cycles consolidation chemotherapy were used:DDP 75mg/m2 D1+docetaxel 75mg/m2 D1, Q3W
  Interventions: Radiation: intensity modulated radiation therapy in both arms; Drug: concurrent chemotherapy with radiation
- standard dose (Active Comparator): concurrent chemoradiation:CT:DDP 25mg/m2 D1+Docetaxel 25mg/m2 D1,Weekly for 5 wks;RT：50Gy/25F/5W(3D-CRT or IMRT).Then,2 cycles consolidation chemotherapy were used:DDP 5mg/m2 D1+Docetaxel75mg/m2 D1, Q3W
  Interventions: Radiation: intensity modulated radiation therapy in both arms; Drug: concurrent chemotherapy with radiation

INTERVENTIONS:
Radiation: intensity modulated radiation therapy in both arms
Drug: concurrent chemotherapy with radiation — docetaxel plus cisplatin were used weekly in both arms

SUMMARY:
Radiation therapy plus concurrent chemotherapy is now the standard therapy for patients with localized carcinoma of the esophagus selected for nonsurgical treatment. The standard radiation dose is 50-50.4Gy/1.8-2.0Gy/F.All of this were based on 2D radiation technology. Entering new century, 3D-CRT or IMRT has used on esophageal cancer. In China,the recommend radiation dose of concurrent chemoradiation was 60Gy. The study is a clinical phase III, randomized trial to compare the different radiation dose(60Gy vs 50Gy) of concurrent chemoradiation using 3D-CRT or IMRT in patients with unresectable esophageal carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytologic diagnosis of esophageal carcinoma
* ECOG performance status 0-1
* Age:18-70 years
* Joined the study voluntarily and signed informed consent form
* Patients must not have received any prior anticancer therapy
* Unresectable disease, or refuse surgery.Stage Ⅰ-ⅣA（AJCC 2009）
* Target lesions can be measured according to RECIST criteria
* No serious system dysfunction and immuno-deficiency, Adequate organ function including the following: Hemoglobin ≥9 g/dL, WBC≥3x109/L, Neutrophils (ANC )≥1.5x109/L, platelet count ≥100x 109/L, TBIL<1.5 x ULN, ALT and AST ≦ 2.5 x ULN, creatinine ≦ 1.5 x ULN
* Use of an effective contraceptive for adults to prevent pregnancy
* Life expectancy of more than 3 months

Exclusion Criteria:

* Multiple carcinomas of the esophagus,
* Biopsy-proven invasion of the tracheobronchial tree or tracheoesophageal fistula,
* Metastatic disease (M1),
* A primary tumor that extended to within 2 cm of the gastroesophageal junction,
* Prior chemotherapy, prior thoracic radiation, surgical resection of the primary tumor,
* Concurrent pregnancy or lactation, history of a second malignancy other than nonmelanoma skin cancer

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2013-08; Primary Completion 2015-08 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | 5 years

SECONDARY OUTCOMES:
Overall survival | 5 years

OTHER OUTCOMES:
local control rate; relapse location; toxicity | 5 years
radiation-related advent events | at least 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Xiao Zheng, MD, Principal Investigator — Zhejiang Cancer Hospital
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China